CLINICAL TRIAL: NCT02890849
Title: Clinical Research for the Consistency Analysis of PD-L1 in Cancer Tissue and Plasma Exosome
Acronym: RadImm01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy Director, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-004
Record Dates: First submitted 2016-08-24; First posted 2016-09-07 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: NSCLC
MeSH Terms: interventions — Liquid Biopsy

ARMS (1):
- a prospective, open, self-controlled phase I clinical study (Experimental): The project is planned to explore the consistency analysis of PD-L1 expression level detected in cancer tissues and pExo.We have designed to detected the expression levels of PD-L1 mRNA and protein in cancer tissue and detected the expression levels of PD-L1 mRNA in pExo.by using variance analysis of repeated measures design information.
  Interventions: Other: Liquid biopsy

INTERVENTIONS:
Other: Liquid biopsy

SUMMARY:
The detection of tissue PD-L1 immunohistochemistry in Non-small cell lung cancer (NSCLC) has an important role in guiding for the treatment of immune detection point. At the same time,tissue detection is time-consuming and laborious, liquid biopsy can reflect the information of tumor tissue,PD-L1 mRNA in plasma exosomes (pExo) is expected to be simple, rapid, non-invasive means of detection. The project is planned to explore the consistency analysis of PD-L1 expression level detected in cancer tissues and pExo.We have designed to detected the expression levels of PD-L1 mRNA and protein in cancer tissue and detected the expression levels of PD-L1 mRNA in pExo.By using variance analysis of repeated measures design information. Thus exploring the consistency analysis of PD-L1 expression level detected in tissues and pExo,guiding clinical practice of radiotherapy combining with immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological histology and/or cytology confirmed malignant tumor;
2. Voluntarily enrolled to participate in,better compliance, cooperate with experimental observations, and sign informed consent.

Exclusion Criteria:

1. Vital organs (e.g., heart, liver, kidney) have serious dysfunction;
2. Patients with a history of autoimmune disease;
3. Patients with participating in other clinical trials at the same time;
4. Other cases that researchers believe that patients should not participate in the present trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10; Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
The match rate of PD-L1 protein expression in cancer tissue and PD-L1 mRNA expression in pExo. | up to one and a half years

SECONDARY OUTCOMES:
The match rate of PD-L1 protein expression and PD-L1 mRNA in tumor tissue. | up to one and a half years

OTHER OUTCOMES:
Correlation between PD-L1 mRNA expression in pExo and immune indexes. | up to one and a half years